CLINICAL TRIAL: NCT03201198
Title: Active for Life: Chronic Obstructive Pulmonary Disease
Acronym: ActiveCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Janet L. Larson, Shaké Ketefian Collegiate Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00119545; R01NR016093 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-06-28 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: physical activity; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Life (Experimental): The Active Life intervention includes structured walking, functional circuit training, stretching and behavior/educational components.
  Interventions: Behavioral: Active Life
- Chair exercises (Sham Comparator): The Chair exercise intervention includes chair exercises, behavioral relaxation and health education.
  Interventions: Behavioral: Chair exercises

INTERVENTIONS:
Behavioral: Active Life — The Active Life intervention focuses on increasing light physical activity (LPA) with 18 sessions over 10 weeks. Each session starts with 20 minutes of walking followed by functional circuit training. The intensity of the exercises and the speed of execution are adjusted to attain a rating of perceived exertion equal to somewhat hard to hard at the end of each circuit. Sessions end with stretching the major muscle groups. Sessions include a behavioral component (self-efficacy enhancing or confidence building) and health education. Subjects are encouraged to increase their total PA by at least 60 minutes a day, focusing on LPA. After completion of the structured intervention subjects will receive 11 5-minute phone coaching sessions and two booster sessions over the next 12 months.
  Arms: Active Life
Behavioral: Chair exercises — Chair exercises focus on toning and stretching from a seated position with 18 sessions over 10 weeks. Each session includes 5 minutes of slow stretching, 20 minutes of faster paced exercises, 5 minutes of slower paced stretches, followed by 5-10 minutes of massage and imagery. Guided imagery is used to promote relaxation. Health education includes topics of interest to people with COPD such as basic lung physiology, pathophysiology of COPD, commonly used medications, breathing techniques, healthy eating and physical activity, relaxation, travel considerations, and energy conservation. After completion of the structured intervention subjects will receive 11 5-minute phone coaching sessions and two booster sessions over the next 12 months.
  Arms: Chair exercises

SUMMARY:
This study examines the effects of an exercise and behavioral program, called Active-Life, to promote physical activity in people with chronic obstructive pulmonary disease. A sedentary lifestyle is very common in older people with chronic disease and if this program is successful it will be used to promote physical activity and improve the health of people with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Physical inactivity is a growing health problem in the United States, especially for older people with chronic diseases such as COPD; in fact people with COPD are among the least active. Low levels of physical activity (PA) are associated with negative health outcomes including an increase in mortality and COPD exacerbations. Current PA guidelines focus on moderate-to-vigorous physical activities (MVPAs) that are too strenuous and not feasible for long term maintenance in many people with COPD. The investigators propose a new paradigm for promoting PA in this population; focus on increasing time spent in light physical activity (LPA) and decreasing time spent in sedentary behavior. Growing evidence suggests that substantial health benefits are associated with increases in the volume of LPA. The investigators are testing the efficacy of the Active-for-Life (Active-Life) intervention. The central hypothesis is that Active-Life will have positive effects on objectively measured PA. Active-Life is a 10 week intervention designed to increase total PA with an emphasis on increasing the time spent in LPA and decreasing sedentary time. Active-Life establishes a goal for subjects, to increase total PA, combined LPA and MVPA, at least 60 minutes a day. This far exceeds the effects of other published PA interventions for people with COPD and if successful will advance PA science in clinically important ways. The Active-Life program was developed by Dr. Larson and through a series of preliminary studies; its feasibility is well established and preliminary data are promising. The investigators are conducting a randomized controlled trial comparing Active-Life against an active control. They will enroll 183 people with moderate to very severe COPD. Outcomes will be measured at baseline, end of the 10 week intervention and at 3, 6 and 12 months after the end of the intervention. The primary dependent variables are objectively measured PA and sedentary behavior, measured with ActivPAL and Actigraph accelerometers simultaneously. Secondary outcome measures are indicators of frailty: 6-minute distance walk, isometric strength of knee flexors and extensors, Short Physical Performance Battery and self-reported physical function. Potential mediators include barriers-efficacy for PA and outcome expectations for PA.

ELIGIBILITY:
Inclusion Criteria:

* No acute exacerbations or major illnesses requiring hospitalization in the last 8 weeks.
* No history of other major lung diseases as primary pulmonary problem, history of a recent heart attack or recent onset of chest pains with activity or increasing episodes of chest pain (unstable angina).
* No other health problems or mobility problems that limit physical activity.
* Sedentary (less than 30 minutes of moderate activity 3 days/week)

Exclusion Criteria:

* Acute exacerbations or major illnesses requiring hospitalization in the last 8 weeks.
* History of other major lung diseases as primary pulmonary problem, history of a recent heart attack or recent onset of chest pains with activity or increasing episodes of chest pain (unstable angina).
* Other health problems or mobility problems that limit physical activity.
* Participated in a structured exercise program or pulmonary rehabilitation within the last year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Larson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
At this point the investigators have no plans to share IPD, but would consider a request to share deidentified data if it had the potential to advance science in the promotion of physical activity for older adults

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects recruited had a diagnosis of COPD, were between the ages of 60-85 years, and had an FEV1%predicted less than 80%. Subjects recruited were stratified by gender and FEV1%predicted severity as part of the randomization process.
Pre-assignment Details: A total of 182 subjects were enrolled and randomized across both groups. Five subjects were not able to complete baseline assessment leaving 177 randomized subjects who completed baseline assessment.
Period: Overall Study
Arm/Group | Active Life | Chair Exercises
Started | 92 | 90
Completed | 55 | 50
Not Completed | 37 | 40
Not completed — Did not complete f reasons; lost to follow-up, subject withdrew, family illnesses, moving, etc. | 35 | 37
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Life | Chair Exercises | Total
Number analyzed (Participants) | 92 | 90 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was collected at the time of baseline spirometry. A total of 11 subjects did not have baseline spirometry completed. Eight subjects in the treatment arm and 3 subjects in the control arm did not have age reported at baseline assessment.
  years
    number analyzed (Participants) | 82 | 84 | 166
    (all) | 68.5 (7.8) | 70.3 (8.5) | 69.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender was not reported in 11 subjects during baseline spirometry. 8 subjects in the treatment arm and 3 subjects in the control arm
  Participants
    number analyzed (Participants) | 82 | 84 | 166
    Female | 37 | 38 | 75
    Male | 45 | 46 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race not recorded for 12 subjects at baseline. 5 participants did not complete baseline assessments. 17 total unknown
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 1 | 2 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 13 | 22
    White | 70 | 68 | 138
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 10 | 7 | 17
FEV1%Predicted [Mean (Standard Deviation); unit: Percent of actual to predicted] — Population: Eleven subjects (8 in treatment arm, 3 in control arm) did not report baseline spirometry
  Percent of actual to predicted
    number analyzed (Participants) | 82 | 84 | 166
    (all) | 53.77 (15.6) | 56.99 (13.5) | 55.4 (14.5)

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Physical Activity as Measured by Upright Time (Minutes Per Day) Monitored by ActivPal Monitor
Description: The primary dependent variables are the time spent in physical activity (PA) as measured by Upright time monitored in each of the five intervals of the study over a 15-month period. PA will be measured for 7 consecutive days at each measurement using the ActivPal monitor. Each subject must have at least 4 of 7 valid monitoring days in each monitored period. The monitored periods are: baseline (T1), immediate post-intervention (T2), 3-month follow-up post intervention (T3), 6 month follow-up (T4), 12 month follow-up period (T5)
Time Frame: 7 days of continuous activity monitoring w as monitored on each participants at each of five test periods (T1-T5)
Population: Number of participants who were analyzed at each time period (T1-T5) varied due to participants withdrawing, not being available to keep their test appointments, illness, etc. T1=baseline, T2=testing at completion of intervention, T3= 3 months following intervention, T4=6 months following intervention, T5=12 months following intervention
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Active Life | Chair Exercises
Number analyzed (Participants) | 90 | 87
minutes per day
  Baseline-T1: number analyzed (Participants) | 71 | 78
  Baseline-T1 | 278 (144) | 269 (138)
  T2: number analyzed (Participants) | 54 | 45
  T2 | 293 (138) | 285 (130)
  T3: number analyzed (Participants) | 53 | 44
  T3 | 293 (156) | 279 (138)
  T4: number analyzed (Participants) | 52 | 48
  T4 | 282 (154) | 257 (99)
  T5: number analyzed (Participants) | 50 | 41
  T5 | 277 (145) | 299 (146)

2. Primary Outcome: Time Spent in Sedentary Behavior
Description: The primary dependent variable are the time spent in sedentary activity as measured as Sedentary Activity (SA) time monitored in each of the five intervals of the study over a 15-month period. SA will be measured for 7 consecutive days at each interval using the ActivPal monitor. Each subject must have at least 4 of 7 valid monitoring days in each monitored period. The monitored periods are: baseline (T1), immediate post-intervention (T2), 3-month follow-up post intervention (T3), 6 month follow-up (T4), 12 month follow-up period (T5)
Time Frame: 7 days of continuous activity monitoring at each interval
Population: Participant/unit totals differ from overall number analyzed due to invalid or incomplete monitoring of subjects or subjects withdrawals between intervals.
Measure: Mean (Standard Deviation); unit: average minutes per day
Arm/Group | Active Life | Chair Exercises
Number analyzed (Participants) | 90 | 87
average minutes per day
  Baseline (T1): number analyzed (Participants) | 71 | 78
  Baseline (T1) | 683 (180) | 698 (187)
  T2: number analyzed (Participants) | 54 | 45
  T2 | 661 (173) | 658 (177)
  T3: number analyzed (Participants) | 53 | 44
  T3 | 661 (180) | 672 (180)
  T4: number analyzed (Participants) | 52 | 48
  T4 | 683 (182) | 681 (160)
  T5: number analyzed (Participants) | 50 | 41
  T5 | 671 (174) | 639 (169)

3. Secondary Outcome: Six-minute Walk Test
Description: This is the maximal distance a subject can walk during six minutes.
Time Frame: Measured at baseline, end of 10 week intervention and at 3, 6, and 12 months after the completion of the 10 week intervention
Population: Participant/unit totals differ from overall number analyzed due to invalid or incomplete testing of subjects or subjects withdrawals between intervals.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Active Life | Chair Exercises
Number analyzed (Participants) | 90 | 87
Feet
  Baseline (T1): number analyzed (Participants) | 70 | 80
  Baseline (T1) | 1241 (306) | 1202 (324)
  T2: number analyzed (Participants) | 54 | 52
  T2 | 1368 (254) | 1234 (339)
  T3: number analyzed (Participants) | 52 | 47
  T3 | 1320 (343) | 1281 (295)
  T4: number analyzed (Participants) | 49 | 47
  T4 | 1339 (280) | 1272 (294)
  T5: number analyzed (Participants) | 49 | 87
  T5 | 1311 (267) | 1264 (307)

ADVERSE EVENTS:
Time Frame: 15 months for each subject enrolled who completed the entire study period
Arm/Group | Active Life | Chair Exercises
All-Cause Mortality (participants affected / at risk) | 4/82 | 1/84
Serious Adverse Events (participants affected / at risk) | 7/82 | 5/84
Other Adverse Events (participants affected / at risk) | 17/82 | 12/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Life (N=82) | Chair Exercises (N=84)
acute exacerbation requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) — Acute exacerbation of underlying condition (COPD) requiring hospitalization while subject was enrolled in clinical trial
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Life (N=82) | Chair Exercises (N=84)
Exercise intolerance due to pain or injury, non-serious (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Fall with non-serious injury (Injury, poisoning and procedural complications) | 11 (11) | 7 (7) — Fall from any cause, not necessarily related to enrollment in study

LIMITATIONS AND CAVEATS:
Limitations include decreased recruitment in non-white populations. Attempts were made to recruit from minority groups but not successful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT03201198/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03201198/ICF_001.pdf